CLINICAL TRIAL: NCT04028388
Title: A Multicentre Phase 2b Trial to Evaluate the Efficacy and Tolerability of ModraDoc006/r in Subjects With Metastatic Castration Resistant Prostate Cancer (mCRPC), Suitable for Treatment With a Taxane
Brief Title: ModraDoc006/r vs Docetaxel IV in Metastatic Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Modra Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M18MDP
Record Dates: First submitted 2019-07-17; First posted 2019-07-22 (Actual); Results first posted 2024-04-17 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-01

CONDITIONS: Prostate Cancer Metastatic; Castration-resistant Prostate Cancer
MeSH Terms: interventions — Docetaxel; Injections

STUDY DESIGN:
Intervention Model Description: One-hundred RECIST 1.1 evaluable patients will be randomized 1:1 to treatment with ModraDoc006/r versus standard i.v. docetaxel. The treatment outcome will be estimated and used as the basis for the design of the future pivotal phase 3 trial. The sample size of 50 evaluable patients per cohort will provide a sufficiently precise point estimate of the primary endpoint radiographic Progression Free Survival (rPFS) in both groups to calculate the sample size for the pivotal study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Docetaxel IV (Active Comparator): This study arm will receive docetaxel at 75 mg/m2 given i.v. as a one-hour infusion on day 1 every 21 days plus 5 mg oral prednisone twice daily.
  Interventions: Drug: Docetaxel in Parenteral Dosage Form
- ModraDoc006/r (Experimental): This cohort will receive ModraDoc006/r 30 mg oral docetaxel in combination with 200 mg ritonavir in the morning and 20 mg oral docetaxel in combination with 100 mg ritonavir in the evening (7-12 hours after the morning dose), on Day 1, 8 and 15 of a 21-day cycle, plus 5 mg oral prednisone twice daily.
  Interventions: Drug: ModraDoc006/r

INTERVENTIONS:
Drug: Docetaxel in Parenteral Dosage Form — Treatment with IV docetaxel at 75 mg/m2 given as a one-hour infusion on day 1 every 21 days plus 5 mg oral prednisone twice daily
  Other Names: Taxotere
  Arms: Docetaxel IV
Drug: ModraDoc006/r — Treatment with twice daily once weekly (BIDW) ModraDoc006 (oral docetaxel) 10mg tablets in combination with ritonavir 100mg tablets
  Other Names: oral docetaxel formulation
  Arms: ModraDoc006/r

SUMMARY:
This is a multicenter phase 2b study to evaluate the efficacy and tolerability of ModraDoc006 in combination with ritonavir (denoted ModraDoc006/r) in patients with metastatic castration-resistant prostate cancer, suitable for treatment with a taxane.

DETAILED DESCRIPTION:
This is an open label 1:1 randomized Phase 2b trial to determine the efficacy and tolerability of oral ModraDoc006/r versus i.v. docetaxel in mCRPC subjects. Cohort 1 will receive i.v. docetaxel at 75 mg/m2 every 3 weeks (Q3W). Cohort 2 will receive 30 mg ModraDoc006 in combination with 200 mg ritonavir in the morning and 20 mg ModraDoc006 in combination with 100 mg ritonavir in the evening (7-12 hours after the morning dose), on Day 1, 8 and 15 of a 21-day cycle (BIDW). All patients will also receive 5 mg oral prednisone twice daily. Treatment in both cohorts will continue until disease progression, unacceptable toxicity, or discontinuation for any other reason. The end of the trial is defined as the time point when all subjects have discontinued trial treatment and have been given follow-up for safety measurements according to the trial assessment schedule.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Histologically or cytologically proven prostate cancer with evidence of progressive mCRPC, defined as:

   1. Castrate levels of testosterone, defined as ≤ 50 ng/dL (or ≤ 0.50 ng/mL or 1.73 nmol/L)
   2. Evidence of progressive metastatic disease as defined by radiographic disease progression or Prostate Specific Antigen (PSA) progression
   3. With an indication for systemic treatment with docetaxel according to the standard of care
3. Measurable tumour lesions, defined as pelvic and/or extra-pelvic nodal lesions ≥1.5 cm in the short axis or visceral lesions ≥1.0 cm in the longest dimensions and measurable according to RECIST v1.1, bone metastasis as evaluated with 99mTc-methylene diphosphonate (MDP) radionuclide bone scintigraphy
4. Resolution of toxicity of prior therapy to < grade 2 (except for alopecia), as defined by CTCAE v5.0
5. Adequate haematological, renal and hepatic functions:

   1. Hemoglobin ≥ 6.0 mmol/l (>9.6 g/dL)
   2. Absolute Neutrophil Count (ANC) ≥ 1.5 x 109 /L
   3. Platelet count ≥ 100 x 109 /L
   4. Hepatic function defined by serum bilirubin ≤ Upper Limit of Normal (ULN), Alanine Amino Transferase (ALAT) and Aspartate Amino Transferase (ASAT) ≤ 1.5 x ULN concomitant with alkaline phosphatase ≤ 2.5 × ULN.
   5. Renal function defined by serum creatinine ≤ 1.5 x ULN or creatinine clearance ≥ 50 ml/min (by Cockcroft-Gault formula, or MDRD).
6. World Health Organisation Performance Status (WHO-PS) of 0-2
7. Estimated life expectancy of at least 12 weeks
8. Able and willing to swallow oral medication
9. Able and willing to undergo radiologic scans (CT scan)
10. Able and willing to give written informed consent according to local guidelines

Exclusion Criteria:

1. Any treatment with investigational drugs, chemotherapy or immunotherapy within 4 weeks prior to receiving the first dose of investigational treatment. Palliative radiotherapy (1x8 Gy dose) is allowed before and during the study, but not in the week prior to start of study treatment.
2. Subjects who have had prior treatment with taxanes.
3. Subjects with symptomatic brain metastases. Subjects asymptomatic in the absence of corticosteroids and anticonvulsant therapy for ≥6 weeks are eligible. Radiotherapy for brain metastasis must have been completed ≥6 weeks prior to start of trial. Brain metastasis must be stable with verification by imaging (e.g. brain MRI or CT completed at screening, demonstrating no current evidence of progressive brain metastases). Subjects are not permitted to receive anti-epileptic drugs or corticosteroid treatment indicated for brain metastasis. Subjects with a history of leptomeningeal metastases are not eligible.
4. Current malignancies other than mCRPC with exception of adequately treated basal or squamous cell carcinoma of the skin, or adequately treated non-muscular invasive bladder cancer.
5. Absence of highly effective method of contraception as of cycle one day one (C1D1). Men enrolled in this trial must agree to use a highly effective contraceptive method throughout the study.
6. Uncontrolled hypertension (systolic > 150 mm Hg and/or diastolic > 100 mm Hg)
7. Unresolved (>grade 0 as defined by CTCAE version 5.0) gastrointestinal toxicities (pre-existing mucositis, diarrhea or nausea/vomiting)
8. Grade ≥ 2 motor ≥ 2 motor or sensory neuropathy symptoms (as defined by CTCAE version 5.0)
9. Known hypersensitivity to any of the study drugs or excipients or taxanes
10. Concomitant use of P-glycoprotein (P-gp , MDR), Cytochrome P450 (CYP)3A, Organic Anion-Transporting Polypeptide (OATP)1B1, OATP1B3 and Multidrug resistance-associated protein 2 (MRP2) modulating drugs such as Ca+- entry blockers (verapamil, dihydropyridines), cyclosporine, quinidine and grapefruit juice, concomitant use of HIV medications, other protease inhibitors, (non) nucleoside analogues, or St. John's wort
11. Bowel obstruction or motility disorder that may influence the resorption of drugs as judged by the treating physician
12. Major surgical procedures within 21 days prior to providing informed consent
13. Active acute or chronic infection, which is not controlled by appropriate medication (at the discretion of the treating physician)
14. Known positivity for Human Immunodeficiency Virus HIV-1 or HIV-2 type
15. Patients with known active infection of hepatitis B/C (HBC), or E (patients who are anti-HBC positive but HBsAg negative are eligible to participate in this study)
16. Clinically significant (i.e. active) cardiovascular disease defined as stroke, transient ischemic attack (TIA), myocardial infarction, unstable angina, or congestive heart failure within ≤ 6 months prior to first trial treatment
17. Evidence of any other medical conditions (such as treatment-resistant peptic ulcer disease, erosive oesophagitis or gastritis, infectious or inflammatory bowel disease, diverticulitis, or pulmonary embolism within 4 weeks of randomization, or psychiatric illness, drug or alcohol abuse, physical examination or laboratory findings) that may interfere with the planned treatment, affect subject compliance or place the subject at high risk of treatment-related complications
18. Legal incapacity

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2019-07-17 (Actual); Primary Completion 2021-11-29 (Actual); Study Completion 2021-11-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: M Keessen, MSc, MBA, Study Director — Modra Pharmaceuticals
Locations (28):
- United States (4):
  - Karmanos Cancer Institute, Detroit, Michigan
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Providence Cancer Institute, Portland, Oregon
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
- Czechia (2):
  - Nemocnice Liberec, Liberec
  - Urologicke oddeleni FTN, Prague
- Germany (3):
  - Universitätsmedizin Göttingen, Göttingen
  - Studienpraxis Urologie, Nürtingen
  - Universitätsklinikum Tübingen, Tübingen
- Hungary (4):
  - Orszagos Onkologiai Intezet (National Institute of Oncology), Budapest
  - Debreceni Egyetem Klinikai Központ, Debrecen
  - Petz Aladár Megyei Oktató Kórház, Győr
  - Jasz-Nagykun-Szolnok Megyei - Hetenyi Geza Korhaz - Rendelointezet - Onkologiai Kozpont, Szolnok
- Poland (3):
  - Przychodnia Lekarska "KOMED", Konin
  - Instytut Centrum Zdrowia Matki Polki, Lodz
  - Centrum Onkologii - Instytut im. Marii Skłodowskiej-Curie, Warsaw
- Russia (12):
  - Regional State Budgetary Healthcare Institution "Altai regional oncology dispensary", Barnaul
  - Limited Liability Company "EVIMED, Chelyabinsk
  - Regional State Budget Institution "Krasnoyarsk Territorial Clinical Hospital n.a. A.I.Kryzhanovskogo", Krasnoyarsk
  - Federal State Institution "Russian Cancer Research Center named after N. N. Blokhin" RAMS, Moscow
  - CJSC Medical Center "AVICENNA", Novosibirsk
  - Federal state budget institution "National medical research radiological center " of the Ministry of healthcare of the Russian Federation, branch - A. Tsyb Medical Radiological Research Center, Obninsk
  - Clinical Oncological Dispensary of Omsk Region, Omsk
  - Leningrad Region Onco Dispensary, Saint Petersburg
  - Limited Liability Company "Klinika Andros [Andros Clinic]", Saint Petersburg
  - National medical research center of oncology n.a. N.N. Petrov, Saint Petersburg
  - Pavlov First Saint Petersburg State Medical University, Saint Petersburg
  - Sverdlovsk Regional Clinical Hospital No. 1, Yekaterinburg

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The number of enrollment is not equal to the number of patients started, because 32 patients did not meet the inclusion criteria.
Groups:
- Docetaxel IV: In this study arm patients received docetaxel at 75 mg/m2 given i.v. as a one-hour infusion on day 1 every 21 days (Q3W), plus 5 mg oral prednisone twice daily.
  Premedication with dexamethasone was required.
  Docetaxel in Parenteral Dosage Form: Treatment with IV docetaxel at 75 mg/m2 given as a one-hour infusion on day 1 every 21 days plus 5 mg oral prednisone twice daily.
- ModraDoc006/r: In this study arm patients initially received ModraDoc006 30 mg in combination with ritonavir 200 mg in the morning and ModraDoc006 20 mg in combination with 100 mg ritonavir in the afternoon, 7 to 12 hours after the morning dose (=ModraDoc006/r 30-20/200-100 mg) twice daily once weekly (BIDW) on Days 1, 8, and 15 of a 21-day cycle, plus prednisone 5 mg orally twice daily. After a total of 39 patients randomized (21 patients in ModraDoc006/r), the morning dose was amended to 20 mg in combination with ritonavir 200 mg (=ModraDoc006/r 20-20/200-100 mg).
  No dexamethasone premedication was given. ModraDoc006/r: Treatment with twice daily once weekly (BIDW) ModraDoc006 (oral docetaxel) 10mg tablets in combination with ritonavir 100mg tablets.
Period: Overall Study
Arm/Group | Docetaxel IV | ModraDoc006/r
Started | 51 | 52
Completed | 46 | 46
Not Completed | 5 | 6
Not completed — Evaluations missing | 3 | 6
Not completed — Not started | 2 | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics have been provided for the Full Analysis Set (FAS). All patients who received at least 1 dose of intravenous docetaxel (Cohort 1) or 1 full cycle of ModraDoc006/r (Cohort 2) and had at least 1 post-baseline tumor assessment were included in the FAS.
Groups:
- Docetaxel IV: Patients received docetaxel at 75 mg/m2 i.v. Q3W, with dexamethasone premedication, plus 5 mg oral prednisone twice daily.
- ModraDoc006/r: Patients received ModraDoc006/r either at 30-20/200-100 mg or at 20-20/200-100 mg BIDW, plus 5 mg oral prednisone twice daily.
- Total: Total of all reporting groups
Arm/Group | Docetaxel IV | ModraDoc006/r | Total
Number analyzed (Participants) | 46 | 46 | 92
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 11 | 22
  >=65 years | 35 | 35 | 70
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.8 (6.6) | 67.0 (6.9) | 67.4 (6.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 46 | 46 | 92
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 44 | 45 | 89
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 44 | 44 | 88
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Hungary | 7 | 3 | 10
  United States | 11 | 13 | 24
  Czechia | 3 | 2 | 5
  Poland | 3 | 3 | 6
  Germany | 2 | 3 | 5
  Russia | 20 | 22 | 42
ECOG Performance Status at study entry [Count of Participants; unit: Participants]
  Performance status 0 | 17 | 29 | 46
  Performance status 1 | 28 | 15 | 43
  Performance status 2 | 1 | 2 | 3
Time since diagnosis of mCRPC [Mean (Standard Deviation); unit: Months] | 12.24 (14.92) | 15.72 (29.48) | 13.98 (23.30)
RECIST measurable disease at study entry [Count of Participants; unit: Participants]
  Yes | 33 | 36 | 69
  No | 13 | 10 | 23

OUTCOME MEASURES:

1. Primary Outcome: Radiographic Progression Free Survival (rPFS)
Description: Evaluation of rPFS that will be observed as measured by Prostate Cancer Clinical Trials Working Group 3 (PCWG3) criteria, in patients with metastatic prostate cancer after treatment with ModraDoc006/r or docetaxel IV.
  Radiographic disease progression was defined by the local assessment of:
  * Progressive disease by RECIST v1.1. for soft tissue disease
  * Or the appearance of 2 or more new bone lesions on bone scan (PCWG3)
Time Frame: Time from the date of randomization to the date of the first radiologic progression (per PCWG3 criteria) or death from any cause, whichever occurred first, an average of 1 year.
Population: All patients who received at least 1 dose of intravenous docetaxel (Cohort 1) or 1 full cycle of ModraDoc006/r (Cohort 2) and had at least 1 post-baseline tumor assessment were included in the Full Analysis Set (FAS). All patients with an rPFS event.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Docetaxel IV | ModraDoc006/r
Number analyzed (Participants) | 13 | 13
Months | 11.1 [7.9 to 13.1] | 9.5 [6.8 to NA] — The upper limit of the 95% confidence interval was not calculable due to an insufficient number of participants with events.
Statistical Analysis 1: Comparison: Docetaxel IV vs ModraDoc006/r; Test type: Superiority; p = 0.1465, Wilcoxon (Mann-Whitney); Hazard Ratio (HR) = 1.22, 95% CI 2-sided [0.56 to 2.65]

2. Secondary Outcome: Adverse Event Profile (Safety)
Description: The hematological and non-hematological safety profile of ModraDoc006/r will be assessed by clinical and laboratory evaluations according to CTCAE v5.0.
Time Frame: Evaluation of all adverse events during the complete study treatment until 28 days after the last intake, an average of 1 year.
Population: The Safety Population (SAF) was used for the evaluation of safety. All patients receiving at least 1 dose of trial medication in either study arm were included in the SAF.
Measure: Count of Participants; unit: Participants
Arm/Group | Docetaxel IV | ModraDoc006/r
Number analyzed (Participants) | 49 | 52
Participants
  Any adverse event | 48 | 50
  Any treatment-related adverse event | 43 | 43
  Adverse events leading to treatment discontinuation | 12 | 13
  Serious adverse events | 16 | 13
  Treatment-related serious adverse events | 8 | 6
  Serious adverse events leading to death | 3 | 3
  Treatment-related serious adverse events leading to death | 0 | 2
  Serious adverse events leading to treatment discontinuation | 5 | 5

3. Secondary Outcome: Overall Response Rate (ORR)
Description: Percentage of patients evaluable for radiological response (ERR) per Prostate Cancer Working Group 3 (PCWG3)-modified Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by CT/MRI with best overall response of either Complete Response (CR), i.e. disappearance of all target lesions, or Partial Response (PR), i.e. ≥30% decrease in the sum of the longest diameter of target lesions. PCGW3-modified RECIST 1.1 criteria implements the requirement for confirmation of progression at least 6 weeks later for bone lesions at all measurement time points, and for soft tissue lesions after the first measurement (after 2 months) only. Tumor measurements were scheduled after every 8 treatment weeks for the first 24 weeks (i.e. during Week 9, Week 17 and Week 25) and every 12 weeks thereafter.
Time Frame: From baseline during the complete study treatment, including follow-up visit 28 days after the last treatment, an average of 1 year.
Population: Population evaluable for radiological response (ERR). Patients with measurable lesions according to RECIST v1.1, that have received at least 6 weekly administrations of ModraDoc006/r or 2 standard three-weekly cycles of i.v. docetaxel were included. Response was evaluated according to RECIST v1.1 and PCWG3 criteria.
Measure: Number (95% Confidence Interval); unit: Percentage of participants analyzed
Arm/Group | Docetaxel IV | ModraDoc006/r
Number analyzed (Participants) | 31 | 34
Percentage of participants analyzed | 38.7 [21.8 to 57.8] | 44.1 [27.2 to 62.1]

4. Secondary Outcome: Disease Control Rate (DCR)
Description: Disease control rate is calculated by the percentage of patients with Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), ≥30% decrease in the sum of the longest diameter of target lesions; and Stable Disease (SD), ≤20% increase to <30% decrease in the sum of the longest diameter of target lesions per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by CT/MRI. Disease control rate is presented by treatment group for patients that were evaluable for radiological response for the overall study.
Time Frame: From baseline through study completion, an average of 1 year
Population: Population evaluable for radiological response (ERR).
Measure: Number (95% Confidence Interval); unit: Percentage of participants analyzed
Arm/Group | Docetaxel IV | ModraDoc006/r
Number analyzed (Participants) | 31 | 34
Percentage of participants analyzed | 96.8 [83.3 to 99.9] | 88.2 [72.5 to 96.7]

5. Secondary Outcome: Duration of Response (DOR)
Description: DOR is defined as the median time in months from documentation of first tumor response to the first objective evidence of radiologic progression, as measured per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by CT/MRI, in the subpopulation of patients experiencing a Complete Response (CR), i.e. Disappearance of all target lesions; and Partial Response (PR), i.e. ≥30% decrease in the sum of the longest diameter of target lesions.
Time Frame: From baseline through study completion, an average of 1 year
Population: Population evaluable for radiological response (ERR).
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Docetaxel IV | ModraDoc006/r
Number analyzed (Participants) | 31 | 34
Months | NA [1.5 to NA] — The median months in Docetaxel IV was not estimable due to an insufficient number of participants with events. The upper limit of the 95% confidence interval was not calculable due to an insufficient number of participants with events. | 4.9 [1.6 to NA] — The upper limit of the 95% confidence interval was not calculable due to an insufficient number of participants with events.
Statistical Analysis 1: Comparison: Docetaxel IV vs ModraDoc006/r; DOR is calculated in the subpopulation of subjects experiencing a response (CR or PR). Hazard Ratio < 1 means that tested drug (ModraDoc006/r) has better outcome; Test type: Superiority; p = 0.4576, Log Rank; Hazard Ratio (HR) = 1.76, 95% CI 2-sided [0.39 to 7.93]

6. Secondary Outcome: Time to Progression (TTP)
Description: Time to Progression is defined as the time from the date of randomization to the date of the first radiologic progression per PCWG3 criteria.
Time Frame: Time from the date of randomization to the date of the first radiologic progression, an average of 1 year.
Population: Full Analysis Set
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Docetaxel IV | ModraDoc006/r
Number analyzed (Participants) | 46 | 46
Months | 11.1 [8.4 to NA] — The upper limit of the 95% confidence interval was not calculable due to an insufficient number of participants with events. | NA [6.8 to NA] — The median months in ModraDoc006/r was not estimable due to an insufficient number of participants with events. The upper limit of the 95% confidence interval was not calculable due to an insufficient number of participants with events.
Statistical Analysis 1: Comparison: Docetaxel IV vs ModraDoc006/r; Difference between the cohorts is tested with Log-rank test and estimated using Univariate Cox model. Wilcoxon test is used if proportional hazards assumption is not fulfilled. Hazard Ratio < 1 means that tested drug (ModraDoc006/r) has better outcome; Test type: Superiority; p = 0.0776, Wilcoxon (Mann-Whitney); Hazard Ratio (HR) = 1.5, 95% CI 2-sided [0.65 to 3.48]

7. Secondary Outcome: PSA Response Rate
Description: PSA decline of >50% from baseline with confirmatory read ≥3 weeks later, based on the Prostate Cancer Working Group 3 (PCWG3) criteria recommendations.
Time Frame: From baseline through study completion, an average of 1 year
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Docetaxel IV | ModraDoc006/r
Number analyzed (Participants) | 46 | 46
Participants | 26 | 23

8. Secondary Outcome: PSA-PFS
Description: Prostate-Specific Antigen Progression-Free Survival (PSA-PFS) according to Prostate Cancer Working Group 3 (PCWG3) guidance.
  Prostate-specific antigen progression was defined as per PCWG3 guidance:
  * If a patient presented first a decline from baseline, progression was defined as the first PSA increase that was ≥25% and ≥2 ng/mL above the nadir, and which was confirmed by a consecutive second value ≥3 weeks later that fulfilled the same criteria (i.e., a confirmed rising trend)
  * If a patient did not present a decline from baseline, progression was defined as the first PSA increase that was ≥25% and ≥2 ng/mL increased from baseline beyond 12 weeks.
Time Frame: Time from the date of randomization to the date of the first prostate-specific antigen progression or death from any cause, whichever occurred first, an average of 1 year.
Population: Full Analysis Set
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Docetaxel IV | ModraDoc006/r
Number analyzed (Participants) | 46 | 46
Months | 7.7 [4.9 to 11.3] | 4.9 [3.5 to 7.6]
Statistical Analysis 1: Comparison: Docetaxel IV vs ModraDoc006/r; [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p = 0.2539, Log Rank; Hazard Ratio (HR) = 1.4, 95% CI 2-sided [0.79 to 2.49]

9. Secondary Outcome: Time to PSA Progression
Description: Time to PSA progression was defined as the time from the date of randomization to the PSA progression as defined by Prostate Cancer Working Group 3 (PCWG3).
  Prostate-specific antigen progression was defined as per PCWG3 guidance:
  * If a patient presented first a decline from baseline, progression was defined as the first PSA increase that was ≥25% and ≥2 ng/mL above the nadir, and which was confirmed by a consecutive second value ≥3 weeks later that fulfilled the same criteria (i.e., a confirmed rising trend)
  * If a patient did not present a decline from baseline, progression was defined as the first PSA increase that was ≥25% and ≥2 ng/mL increased from baseline beyond 12 weeks.
Time Frame: From baseline through study completion, an average of 1 year
Population: Full Analysis Set
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Docetaxel IV | ModraDoc006/r
Number analyzed (Participants) | 46 | 46
Months | 7.7 [4.9 to 11.3] | 4.9 [3.5 to 7.6]
Statistical Analysis 1: Comparison: Docetaxel IV vs ModraDoc006/r; [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p = 0.3062, Wilcoxon (Mann-Whitney); Hazard Ratio (HR) = 1.35, 95% CI 2-sided [0.76 to 2.42]

10. Secondary Outcome: Number of Participants Who Experienced a First Skeletal-Related Event
Description: Number of Participants who Experienced a first Skeletal-Related Event (SRE), i.e. the occurrence of the first skeletal-related event (i.e. radiation therapy or surgery to bone, clinically apparent pathological bone fracture, spinal cord compression, or change of antineoplastic therapy to treat bone pain); from the time of randomisation to the first occurrence.
  Note: Due to small number of SREs the median time to SRE was not evaluable in this patient population.
Time Frame: From baseline through study completion, an average of 1 year
Population: Full Analysis Set
Measure: Number; unit: participants
Arm/Group | Docetaxel IV | ModraDoc006/r
Number analyzed (Participants) | 46 | 46
participants
  Event | 2 | 0
  Censored | 44 | 46

11. Other Pre Specified Outcome: Overall Health-Related Quality of Life Response
Description: An overall Health-Related Quality of Life (HRQoL) improvement was defined by a 10-point or greater increase (= lower score) in the Functional Assessment of Cancer Therapy-global (FACT-G) total score assessment at a post-baseline assessment compared with baseline, at least once during the study.
  The FACT-G questionnaire contains 27-items to measure four domains of HRQoL on a 5 point Likert-type scale in cancer patients: Physical Well-Being (7 items; score range 0-28), Social/Family Well-Being (7 items; score range 0-28), Emotional Well-Being (6 items; score range 0-24), Functional Well-Being (7 items; score range 0-28). Higher scores and increases from baseline indicate higher quality of life.
Time Frame: From baseline through to end of Cycle 10 (each cycle was 21 days)
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Docetaxel IV | ModraDoc006/r
Number analyzed (Participants) | 46 | 46
Participants | 15 | 15

12. Other Pre Specified Outcome: Summary of Improvement by Individual Health- Related Quality of Life Domains
Description: Improvement for individual patients in Health-Related Quality of Life (HRQoL) domains was defined by a ≥3-point increase in the score of a 5 point Likert-like scale at a post-baseline assessment compared with baseline, at least once during study for Functional Assessment of Cancer Therapy (FACT)-G, -P and -T. Improvement was derived using all assessments collected per protocol schedule, i.e. Baseline, End of Cycle 3, 6 and 10 (or End of Treatment if sooner). Higher scores represent better HRQoL.
  FACT-G = global scale, measures four domains of HRQoL in cancer patients: Physical Well-Being (7 items; score range 0-28), Social/Family Well-Being (7 items; range 0-28), Emotional Well-Being (6 items; range 0-24), Functional Well-Being (7 items; range 0-28). Total score (range 0-108) FACT-P = prostate cancer sub scale (12 items; score range 0-48). Total score (FACT-G total score + FACT-P), range 0-156) FACT-T = taxane specific domain score (16 items, range 0 to 64), Total score (0-172)
Time Frame: Improvement assessed at any timepoint from baseline through to End of Cycle 10 (each cycle was 21 days)
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Docetaxel IV | ModraDoc006/r
Number analyzed (Participants) | 46 | 46
Participants
  ≥3 for FACT-G physical well-being | 9 | 13
  ≥3 for FACT-G social or family well being | 16 | 16
  ≥3 for FACT-G emotional well-being | 23 | 18
  ≥3 for FACT-G functional well-being | 18 | 21
  ≥3 for FACT-P | 21 | 23
  ≥3 for FACT-T specific items | 19 | 23

13. Other Pre Specified Outcome: Overall Health-Related Utility
Description: Mean change from baseline to the End of Cycle 10 in the European Quality of Life Dimension-Five Level Scale (EQD5) is presented.
  For the EQD5, mobility, self-care, usual activities, pain/discomfort, and anxiety/depression were scored on a 5-point scale: no problems (1), slight problems (2), moderate problems (3), severe problems (4), and extreme problems (5). Lower scores and decreases from baseline indicate improved quality of life.
  A visual analog scale (VAS) was used for the patient to evaluate their health state at a particular visit; the scale was numbered from 0 (representing the worst health imaginable) to 100 (representing the best health imaginable), higher scores and increases from baseline indicate improved health.
Time Frame: Assessed from baseline to End of Cycle 10 (each cycle was 21 days)
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: Change of score on a scale
Arm/Group | Docetaxel IV | ModraDoc006/r
Number analyzed (Participants) | 46 | 46
Change of score on a scale
  Mobility | 0.4 (1.1) | 0.4 (1.0)
  Self-care | 0.3 (1.1) | 0.0 (0.7)
  Usual activities | 0.5 (1.3) | 0.1 (0.9)
  Pain/discomfort | 0.4 (1.3) | 0.1 (0.7)
  Anxiety/depression | 0.0 (0.8) | 0.0 (0.8)
  Health state | -9.4 (22.2) | -5.9 (20.5)

14. Other Pre Specified Outcome: World Health Organization Performance Status (Eastern Cooperative Oncology Group) at End of Treatment
Description: Eastern Cooperative Oncology Group (ECOG) scores at the time of end on treatment visit are presented.
  0 = Normal activity
  1. = Symptoms, but nearly ambulatory
  2. = Symptomatic, but in bed <50% of the day
  3. = Needs to be in bed >50% of the day, but not bedridden
  4. = Unable to get out of bed
  5. = Dead
Time Frame: Score assessed at end of treatment visit (up to 2 years).
Population: Safety population (SAF)
Measure: Count of Participants; unit: Participants
Arm/Group | Docetaxel IV | ModraDoc006/r
Number analyzed (Participants) | 49 | 52
Participants
  ECOG Score 0 | 10 | 17
  ECOG Score 1 | 16 | 13
  ECOG Score 2 | 4 | 3
  ECOG Score 3 | 0 | 1
  ECOG Score 4 | 0 | 0
  ECOG Score 5 | 2 | 1

ADVERSE EVENTS:
Time Frame: The adverse events were monitored and collected from the time the patient gave informed consent and throughout the study until 30 days after the last ModraDoc006/r or intravenous docetaxel administration; an average of 1 year.
Arm/Group | Docetaxel IV | ModraDoc006/r
All-Cause Mortality (participants affected / at risk) | 4/49 | 3/52
Serious Adverse Events (participants affected / at risk) | 16/49 | 13/52
Other Adverse Events (participants affected / at risk) | 32/49 | 37/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Docetaxel IV (N=49) | ModraDoc006/r (N=52)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1)
Death (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Aphasia (Nervous system disorders) | 0 (0) | 1 (1)
Hemiparesis (Nervous system disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dental caries (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Peptic ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Acute hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Corona virus infection (Infections and infestations) | 3 (3) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 1 (1) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia viral (Covid-19) (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Docetaxel IV (N=49) | ModraDoc006/r (N=52)
Aspartate aminotransferase increased (Investigations) | 2 (6) | 10 (13)
Alanine aminotransferase increased (Investigations) | 2 (8) | 9 (12)
Gamma-glutamyltransferase increased (Investigations) | 2 (2) | 7 (13)
Weight decreased (Investigations) | 3 (4) | 5 (5)
Blood lactate dehydrogenase increased (Investigations) | 1 (1) | 3 (3)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 3 (3)
Blood bilirubin increased (Investigations) | 0 (0) | 3 (3)
Dypnoea (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (4)
Anemia (Blood and lymphatic system disorders) | 13 (25) | 11 (12)
Neutropenia (Blood and lymphatic system disorders) | 11 (26) | 3 (3)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 7 (14)
Leukopenia (Blood and lymphatic system disorders) | 6 (12) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 6 (9) | 2 (2)
Headache (Nervous system disorders) | 1 (1) | 5 (6)
Dysgeusia (Nervous system disorders) | 1 (1) | 4 (4)
Hypoaesthesia (Nervous system disorders) | 4 (5) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 3 (6)
Fatigue (General disorders) | 13 (15) | 11 (13)
Oedema peripheral (General disorders) | 6 (7) | 8 (13)
Asthenia (General disorders) | 4 (4) | 7 (9)
Peripheral swelling (General disorders) | 1 (1) | 3 (3)
Extravasation (General disorders) | 3 (4) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 12 (27) | 25 (51)
Nausea (Gastrointestinal disorders) | 9 (10) | 17 (29)
Constipation (Gastrointestinal disorders) | 3 (3) | 5 (5)
Stomatitis (Gastrointestinal disorders) | 4 (13) | 3 (5)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 5 (8)
Cystitis noninfective (Renal and urinary disorders) | 0 (0) | 3 (5)
Alopecia (Skin and subcutaneous tissue disorders) | 21 (22) | 13 (14)
Nail disorder (Skin and subcutaneous tissue disorders) | 4 (5) | 4 (6)
Dry skin (Skin and subcutaneous tissue disorders) | 3 (5) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 4 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 5 (6)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (5)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 (12) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 3 (6) | 7 (9)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 3 (4)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 3 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-03-31): https://cdn.clinicaltrials.gov/large-docs/88/NCT04028388/Prot_000.pdf
  • Statistical Analysis Plan (2021-10-07): https://cdn.clinicaltrials.gov/large-docs/88/NCT04028388/SAP_001.pdf